CLINICAL TRIAL: NCT04041141
Title: A Pilot Study Assessing an Oral Stent Device for Radiation Treatments of Oral Cancers
Brief Title: Oral Stent Device for Radiation Treatments of Oral Cancers
Status: Withdrawn | Type: Observational
Why Stopped: replaced with other study
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mark Langer, Professor of Clinical Radiation Oncology, Indiana University
Other Study IDs: IUSCC-0687
Record Dates: First submitted 2019-07-11; First posted 2019-08-01 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Tongue Tumor; Tongue Cancer
Keywords: tongue tumor; tongue cancer; oral cancer
MeSH Terms: conditions — Tongue Neoplasms; Mouth Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Cancer: Patients receiving curative radiation treatment for an oral cancer.
  Interventions: Diagnostic Test: CT Scan; Device: Experimental Oral Stent Device

INTERVENTIONS:
Diagnostic Test: CT Scan — An additional cone beam CT will be repeated at midcourse of therapy (3rd week) and during the end of therapy (5th week)
Device: Experimental Oral Stent Device — Patients undergoing standard of care planning for head and neck tongue cancer will have a radiation plan of the body imaged via CT scan construction with the experimental oral stent device in place

SUMMARY:
The purpose of this study is to examine that ability of the experimental oral stent device to reduce the volume of mandible receiving >55 Gy by 50%during radiation treatment as assessed duri radiation treatment planning. Patients will have CT scans at three time-points during their standard of care radiation treatment. During these visits patients will receive scans via CT or cone beam CT scan, with both the standard and experimental oral stent devices.

During radiation treatment patients will receive the standard oral stent device.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 year old at the time of informed consent
* Ability to provide written informed consent and HIPAA authorization
* Accepted for curative radiation treatment of a tongue tumor, either intact or postoperatively
* Signed consent to study participation
* No history of bleeding disorder
* Platelets within normal limits (150-450 k/cumm)

Exclusion Criteria:

* History of bleeding disorder
* History of allergy to dental grade material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential patients will be identified in the Oncology outpatient clinics or by referrals from outside physicians at the Indiana University Simon Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
The volume of mandible irradiated to >55 Gy | volume irradiated at Day 0

SECONDARY OUTCOMES:
The position of the fiducial marker | Change in position at Day 0, Week 3, Week 5
  Fiducial coordinate measured (mm) on XYZ on planning CT

CONTACTS AND LOCATIONS:
Overall Officials: Mark Langer, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States